CLINICAL TRIAL: NCT02802774
Title: Immobilization of Postoperative Distal Radius Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough study participants
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016033
Record Dates: First submitted 2016-06-02; First posted 2016-06-16 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Distal Radius Fractures
Keywords: Post-operative treatment
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Plaster Splint (Active Comparator)
  Interventions: Other: Plaster Splint
- Velcro Brace (Active Comparator)
  Interventions: Other: Velcro Brace
- Soft Dressing (Active Comparator)
  Interventions: Other: Soft Dressing

INTERVENTIONS:
Other: Plaster Splint — The custom plaster splint is the historical standard. The surgical incision is dressed with non-stick gauze, 4x4 gauze pads, cotton padding, a plaster splint applied to the palmar surface of the palm and forearm, and then a cloth wrap to keep it all in place. Patients will wear the plaster splint for 2 weeks post-op.
  Arms: Plaster Splint
Other: Velcro Brace — The Velcro wrist brace is a commercially available over-the-counter splint which will initially be fitted over a thin layer of non-stick gauze, 4x4 gauze, and cotton padding. Patients will be asked to wear the brace as much as possible for the first 2 weeks post-op.
  Arms: Velcro Brace
Other: Soft Dressing — Patients in the soft dressing group will have non-stick gauze, 4X4 gauze, cotton padding, and a cloth wrap. It will be the same dressing as the custom splint without the plaster slab. Patients wear the soft dressing for the first three days post-op.
  Arms: Soft Dressing

SUMMARY:
The management of distal radius fractures has been in a state of evolution over the past 30 years. Treatment has become increasingly focused on obtaining a stable, internal construct for quick return to normal, daily activities. With the advent of volar locking plates, the wrist fracture is stable before the patient leaves the operating room. As surgical plate and screw constructs become more stable, the need for casting and splinting may be less.

The presumptive "next step" in operative management of distal radius fractures is to do away with the postoperative splint. A review of the available English language literature failed to reveal any studies evaluating the use of postoperative splinting and patient outcomes.

This prospective, randomized study was designed to investigate the use of temporary plaster splints versus removable over-the-counter splits versus soft dressings for post-operative treatment of extra-articular and intra-articular distal radius fractures. The patients will be followed for 12 months evaluating maintenance of fracture reduction and patient outcomes.

DETAILED DESCRIPTION:
A prospective study using multiple surgeons at multiple centers (Community Regional Medical Center and Sierra Pacific Orthopaedic Center) investigating post-operative management of extra and intra articular distal radius fractures treated with volar locking plates. Post-operative management for 2 weeks immediately following surgery will consist of placing 1/3 of patients in a short arm, custom-made, plaster splint, 1/3 with a removable Velcro wrist splint, and 1/3 with a soft dressing. The Velcro wrist brace group will be asked to wear the brace as much as possible during the two weeks and the soft dressing may be removed by the patient on the third day after surgery.

* The custom plaster splint is the historical standard. The surgical incision is dressed with non-stick gauze, 4x4 gauze pads, cotton padding, a plaster splint applied to the palmar surface of the palm and forearm, and then a cloth wrap to keep it all in place.
* The Velcro wrist brace is a commercially available over-the-counter splint which will initially be fitted over a thin layer of non-stick gauze, 4x4 gauze, and cotton padding.
* Patients in the soft dressing group will have non-stick gauze, 4x4 gauze, cotton padding, and a cloth wrap. It will be the same dressing as the custom splint without the plaster slab.

Patients will be randomized using REDCap Randomization module after being consented to participate in the study by the primary investigator or sub-investigator. Each investigator will have the option during and/or after surgery to remove the patient from the group they have been randomized into and treat them as they see appropriate. These patients would be documented but removed from the study follow up.

Patient satisfaction will be evaluated subjectively with the PRWE (Patient-Rated Wrist Evaluation) as well as the Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score. Radiographs will be taken at 2, 6, 12, and 24 weeks postoperatively to measure fracture alignment and healing. Patient reported pain level, range of motion, grip, and pinch strength will be recorded at each visit as well as at a final 1 year follow-up visit. Any complication will be noted. All of these visits are part of the standard of care. The only additional part of their visit would be the brief survey including the QuickDASH and PRWE that they complete with an orthopaedic surgery resident during their visit. In addition at the first follow up appointment at 2 weeks post-surgery, patients will be asked about their satisfaction with the mobility of their wrist and those in the Velcro brace will be asked how often they wore the brace. All data will be collected on a data collection sheet and then entered into a database

ELIGIBILITY:
Inclusion Criteria:

* extra and intra articular distal radius fractures treated with distal locking plates

Exclusion Criteria:

* patients with additional injuries to the ipsilateral wrist such as, distal radial ulnar joint (DRUJ) instability and associated unstable ulna fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation | 24 weeks
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score | 24 weeks
Pain Scale (on a scale from 1-10) | 24 weeks
Grip Strength measured in kilograms | 24 weeks
Pinch Strength measured in kilograms | 24 weeks
Range of Motion measured in degrees | 24 weeks
Radiographic evidence of healing | 24 weeks
  Do the x-rays show evidence of bone healing? Yes/No
Complications that required further medical attention | 24 weeks
  Were there any complications that required further medical attention within the first 6 month after surgery?

SECONDARY OUTCOMES:
Patient Rated Wrist Evaluation | 2 weeks
Patient Rated Wrist Evaluation | 6 weeks
Patient Rated Wrist Evaluation | 12 weeks
Patient Rated Wrist Evaluation | 52 weeks
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score | 2 weeks
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score | 6 weeks
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score | 12 weeks
Quick Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) score | 52 weeks
Pain Scale (on a scale from 1-10) | 2 weeks
Pain Scale (on a scale from 1-10) | 6 weeks
Pain Scale (on a scale from 1-10) | 12 weeks
Pain Scale (on a scale from 1-10) | 52 weeks
Radiographic evidence of healing | 2 weeks
  Do the x-rays show evidence of bone healing? Yes/No
Radiographic evidence of healing | 6 weeks
  Do the x-rays show evidence of bone healing? Yes/No
Radiographic evidence of healing | 12 weeks
  Do the x-rays show evidence of bone healing? Yes/No
Complications that required further medical attention | 2 weeks
  Were there any complications that required further medical attention within the first 6 month after surgery?
Complications that required further medical attention | 6 weeks
  Were there any complications that required further medical attention within the first 6 month after surgery?
Complications that required further medical attention | 12 weeks
  Were there any complications that required further medical attention within the first 6 month after surgery?
Complications that required further medical attention | 52 weeks
  Were there any complications that required further medical attention within the first 6 month after surgery?
Range of Motion measured in degrees | 2 weeks
Range of Motion measured in degrees | 6 weeks
Range of Motion measured in degrees | 12 weeks
Range of Motion measured in degrees | 52 weeks
Grip Strength measured in kilograms | 2 weeks
Grip Strength measured in kilograms | 6 weeks
Grip Strength measured in kilograms | 12 weeks
Grip Strength measured in kilograms | 52 weeks
Pinch Strength measured in kilograms | 2 weeks
Pinch Strength measured in kilograms | 6 weeks
Pinch Strength measured in kilograms | 12 weeks
Pinch Strength measured in kilograms | 52 weeks

OTHER OUTCOMES:
Mobility Satisfaction (Extremely, Very, Somewhat, Not at all) | 2

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Hoekzema, MD, Principal Investigator — UCSF - Fresno
Locations (2):
- United States (2):
  - Sierra Pacific Orthopaedic Center, Fresno, California
  - Community Medical Center, Fresno, California

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data.